CLINICAL TRIAL: NCT06915220
Title: ADAPT Micro-Randomized Trial
Acronym: ADAPT MRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Pedja Klasnja, Associate Professor of Information, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00269831; 5R01HL125440-07 (NIH)
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiac Rehabilitation; Physical activity; mobile health intervention
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study uses a micro-randomized trial (MRT) design to optimize the HeartSteps mHealth intervention for physical activity. The following components are macro-randomized:
  1. Activity Suggestions: Randomized twice daily (probability 0.5), averaging one suggestion per day.
  2. Morning Salience Messages: Randomized daily (probability 0.5), averaging one message every other day.
  3. Planning Prompts: Randomized daily (probability 0.5), averaging one prompt every other day.
  The following components are provided without randomization:
  4, Weekly Reflection: Prompts participants each Sunday to reflect on past activity, set goals, and plan for the next week.
  5, Pull Interventions: In-app features like activity dashboards and planning tools.
  6. Ecological Momentary Assessments (EMA): Daily and weekly surveys on psychosocial constructs related to physical activity.
  This plan collects data to optimize intervention timing and content for better engagement and physical activity outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants receive the HeartSteps mHealth intervention for 3 months to support and increase physical activity. Components include:
  1. Activity Suggestions: Push notifications encouraging walks, randomized twice daily (probability 0.5).
  2. Morning Salience Messages: Notifications highlighting positive aspects of activity, randomized daily (probability 0.5).
  3. Planning Prompts: Notifications to plan next day's activity, randomized daily (probability 0.5).
  4. Weekly Reflection: Prompts each Sunday to reflect on past activity, set goals, and plan for the next week.
  5. Pull Interventions: In-app features like activity dashboards and planning tools.
  6. Ecological Momentary Assessments (EMA): Daily and weekly surveys on psychosocial constructs related to physical activity.
  Participants wear a Fitbit Charge tracker to monitor activity, synced to their MyDataHelps account. The intervention aims to optimize engagement and physical activity levels.
  Interventions: Behavioral: mobile health app

INTERVENTIONS:
Behavioral: mobile health app — HeartSteps is an innovative mobile health (mHealth) app designed for cardiac rehabilitation patients. The app features dynamic push notifications, daily and weekly surveys to capture psychosocial data, and an in-app dashboard that provides feedback on activity levels, goal progress, and reminders. Integrated with a Fitbit Charge tracker, HeartSteps emphasizes behavioral changes through engaging features. The intervention is personalized to meet individual needs and preferences, enhancing patient engagement and promoting sustained physical activity.

SUMMARY:
The goal of this study is to collect quantitative and qualitative data that can be used to optimize the HeartSteps mHealth intervention for physical activity. The current version of the intervention is intended to help patients with heart disease increase and maintain their physical activity long-term. To accomplish this goal, a 3-month pilot micro-randomized trial (MRT) will be conducted with 60 patients who are currently completing or have recently completed phase II cardiac rehabilitation (CR).

The core of the study participation is the use of the HeartSteps intervention over the course of 3 months. This includes wearing the Fitbit Charge activity tracker during waking hours and using the HeartSteps intervention to support their efforts to be active. The HeartSteps intervention consists of two sets of intervention components: (1) components intended to improve participants' affective associations with physical activity, including activity suggestions designed to to trigger positive feelings and associate them with being active, and prompts to bring their awareness to intrinsically motivating aspects of being active; and (2) components that target reflective self-regulatory processes, including graphs for self-monitoring, prompts to plan activity, and weekly activity goals. How exactly, and how much, participants will use HeartSteps will not be prescribed since our goal is to understand naturalistic trajectory of engagement with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Must be a patient within the Michigan Medicine clinical system with data available in the electronic health record after January 1, 2020.
* Age > 18
* Owns and is a daily user of an Android or iPhone smartphone with study supported operating software.
* Understands English to enable informed consent, completion of study-related surveys, and compliance with study notifications.
* Will be completing within 30 days or have completed in the last 30 days the cardiac rehabilitation program at Michigan Medicine based on one of the following indications:

  * Coronary artery disease (including acute coronary syndromes and stable angina) following percutaneous coronary intervention (PCI)
  * Coronary artery disease following coronary artery bypass surgery (CABG)]
  * Valve repair or replacement (either surgical or percutaneous)
  * Coronary artery disease or an acute coronary syndrome not requiring revascularization

Exclusion Criteria:

* Orthopedic or neurological condition limiting ability to actively engage in moderate intensity physical activity (e.g., brisk walking)
* Greater than mild cognitive impairment
* Wrist too large to wear an activity tracker comfortably. This will be assessed by asking participants "If they have ever had difficulty wearing a watch in the past due to the band being too small."
* Currently receiving palliative care and/or in hospice care
* Severe valvular stenosis or regurgitation
* Unrevascularized left main coronary artery disease (> 50% obstruction on angiography) or proximal left anterior descending disease (>70% obstruction on angiography).
* Exercise-induced ventricular tachycardia
* Cardiac arrest within the prior 6 months
* New York Heart Association (NYHA) class III or IV heart failure
* Pulmonary arterial hypertension treated with inhaled or intravenous pulmonary hypertension-specific therapy
* Ejection fraction <40%
* Determined to be unsafe for participation in this program as assessed by a clinical nurse or investigative team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Weekly number of minutes of moderate to vigorous physical activity | Baseline, 12 weeks
  The primary outcome of the study is number of weekly minutes of moderate to vigorous physical activity (MVPA), as assessed by the Fitbit Charge 6 activity tracker.
  Primary analysis will assess the difference in MVPA between the baseline week and the last (i.e. 12th) week of the study.

SECONDARY OUTCOMES:
3-hour step count | 12 weeks
  Number of steps, as assessed by the Fitbit Charge 6 activity tracker, measured in the three-hour window following the randomization of activity suggestions.
  This outcome will be assessed after each decision point for the micro-randomized activity suggestions. Each participant will have two decision points per day for the duration of the study.
Daily step count | 12 weeks
  Number of steps per day, assessed by the Fitbit Charge 6 activity tracker.
Affective exercise experiences (AFFEXX) scale | Baseline, 12 weeks
  A validated 36-item self-report instrument that assesses participants' affective associations with physical activity.
  AFFEXX scale will be administered weekly for the duration of the study. The main analysis of this outcome will assess pre-post differences in the AFFEXX score between baseline and 12th week.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided